CLINICAL TRIAL: NCT05113576
Title: Combining Intratumoral Metabolic Heterogeneity and Dissemination Feature (Dmax) on 18F-FDG PET/CT Improves Prognosis Prediction in Diffuse Large B-Cell Lymphoma
Brief Title: Combining Intratumoral Metabolic Heterogeneity and Dissemination Feature (Dmax) on 18F-FDG PET/CT Improves Prognosis Prediction in DLBCL
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-293
Record Dates: First submitted 2021-11-02; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: diffuse large B-cell lymphoma; Positron emission tomography (PET); metabolic heterogeneity; dissemination; metabolic tumor volume
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: patients with DLBCL

SUMMARY:
This retrospective study aimed to investigate the combined prognostic values of intratumoral metabolic heterogeneity (MH), disseminate feature (Dmax) and total metabolic tumor volume (TMTV) by 2-deoxy-2-[18F]fluoro-D-glucose positron emission tomography/computed tomography ([18F]FDG PET/CT), and establish novel nomograms to improve prognosis prediction in diffuse large B-cell lymphoma (DLBCL)

DETAILED DESCRIPTION:
This retrospective study aimed to investigate the combined prognostic values of intratumoral metabolic heterogeneity (MH), disseminate feature (Dmax) and total metabolic tumor volume (TMTV) by 2-deoxy-2-[18F]fluoro-D-glucose positron emission tomography/computed tomography ([18F]FDG PET/CT), and establish novel nomograms to improve prognosis prediction in diffuse large B-cell lymphoma (DLBCL)

Patients would be retrospectively includedin this study.The inclusion criteria included (1) pathologically proven DLBCL; (2) first-line treatment with R-CHOP or R-CHOP-like chemotherapy including R-miniCHOP and R-ECHOP (rituximab, etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin); (3) at least 2 evaluable hypermetabolic lesions on PET/CT;(4) underwent pre-treatment [18F]FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* (1) pathologically proven DLBCL, (2) first-line treatment with R-CHOP or R-CHOP-like chemotherapy including R-miniCHOP and R-ECHOP (rituximab, etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin),(3) at least 2 evaluable hypermetabolic lesions on PET/CT, (4) underwent pre-treatment [18F]FDG PET/CT

Exclusion Criteria:

* (1) patients who had received surgical resection or other treatments before chemotherapy, (2) patients who had coexistent central system lymphoma or other types of malignancies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 132 patients with DLBCL
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
the accuracy of prognosis prediction | Through study completion, about 6 months
  The accuracy of clinical model, PET models and combined model for prediction

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine and PET/CT Center, The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided